CLINICAL TRIAL: NCT06701058
Title: Active MMP-8 in Oral Fluid for the Detection of Oral and Oropharyngeal Cancer
Status: Completed | Type: Observational
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: Karolinska Institutet (Other); University of Helsinki (Other)
Responsible Party: Principal Investigator, Sebastian Ahlstrand, Principal Investigator, Helsinki University Central Hospital
Other Study IDs: TYH2021220
Record Dates: First submitted 2024-11-06; First posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Oropharyngeal Cancers; Biomarker in Early Diagnosis; Oral Cancer , Oral Squamous Cell Carcinoma, Oral Cavity Cancer; Periodontal Diseases
Keywords: aMMP-8; matrix; metalloproteinase; cancer; carcinoma; oral; oropharyngeal; mouthrinse
MeSH Terms: conditions — Oropharyngeal Neoplasms; Mouth Neoplasms; Squamous Cell Carcinoma of Head and Neck; Periodontal Diseases; Neoplasms; Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — Mouth-rinse MMP-8 point-of-care immuno test
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | US Export: No

GROUPS / COHORTS (2):
- Cancer patients: Oral and oropharyngeal cancer patients
- Control patients: Control participants with no history of any type of cancer cancer in the past five years

SUMMARY:
The goal of this observational study is to evaluate whether the active-matrix metalloproteinase-8 (aMMP-8) mouth-rinse test can help detect oral and oropharyngeal cancers. Researchers measured aMMP-8 levels in mouth-rinse samples collected from 77 cancer participants and 50 non-cancer participants in a clinical setting.

The main question this study seeks to answer:

Can the aMMP-8 mouth-rinse test accurately identify and differentiate cancer participants from non-cancer participants in real-time?

DETAILED DESCRIPTION:
The goal of this prospective study is to evaluate whether the active-matrix metalloproteinase-8 (aMMP-8) mouth-rinse test can detect and differentiate 72 oral and oropharyngeal cancers from 50 control participants.

In sampling process patients were asked to pre-rinse with tap water for 30 s. After one-minute wait, they were asked to rinse their mouth 30 s with 5 mL of distilled water provided in the test kit and to spit it out in a sterile measuring cup.

The sample solution were poured into the opening of the test cassette placed on the test system (ORALyzer®) for quantitative results. After obtaining the quantitative results in 5-6 min, the cassette was promptly removed to conduct the qualitative evaluation (Periosafe®).

The expression of aMMP-8 was compared with various factors, including age, sex, smoking status, periodontitis, tumor size, nodal or distal metastases, cancer stage, histological grade, and tumor site. Statistical analysis was performed to evaluate these relationships.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-confirmed oral or oropharyngeal cancer identified by the following International Classification of Diseases (ICD-10) codes: C00-C06, C08-C10, C13, and C32 according to the American Joint Committee on Cancer (AJCC) 8th Edition
* Adult

Exclusion Criteria:

* In-situ cancer
* Previous cancer diagnosis within five years prior to the examination
* Use of tetracyclines at the time of sampling
* Did not follow the manufacturer's instructions prior to the mouth-rinse sample (i.e. brushing teeth before sampling)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study included participants of all ages and genders. All patients were eligible regardless of other medical conditions, except for those with a history of cancer within five years prior to sampling. Cancer patients were selected from a multidisciplinary meeting, and suitable patients were contacted to assess their willingness to participate. Control participants were recruited from the otorhinolaryngology outpatient clinic, where they were being studied and/or treated for other otorhinolaryngology-related conditions
Sampling Method: Non-Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-18 (Actual)

PRIMARY OUTCOMES:
aMMP-8 levels and status in mouth rinse-samples measured utilizing aMMP-8 Point-of-Care Test | Within two hours from initial sample obtained for this study
  aMMP-8 levels were quantitatively measured in real-time using rapid point-of-care (PoC) chairside kits (Periosafe®, Dentognostics GmbH, Solingen, Germany) and a quantitative reader (Oralyzer®, Dentognostics GmbH, Solingen, Germany) to assess mouth-rinse samples from patients with oral and oropharyngeal cancer in comparison to healthy subjects.
  The threshold for a positive quantitative aMMP-8 result is set at 20 ng/ml, with readings of ≥20 ng/ml considered positive and those <19.9 ng/ml considered negative.

CONTACTS AND LOCATIONS:
Overall Officials: Antti Mäkitie, Prof., Study Director — Helsinki University Central Hospital
Locations (1):
- Helsinki University Central Hospital, Helsinki, Uusimaa, Finland

IPD SHARING:
Plan to Share IPD: Yes
The data presented in this study are available on request from the corresponding author. The data are not publicly available due to patient data confidentiality.

REFERENCES:
- [Background] Keskin M, Rintamarttunen J, Gulcicek E, Raisanen IT, Gupta S, Tervahartiala T, Patila T, Sorsa T. A Comparative Analysis of Treatment-Related Changes in the Diagnostic Biomarker Active Metalloproteinase-8 Levels in Patients with Periodontitis. Diagnostics (Basel). 2023 Feb 27;13(5):903. doi: 10.3390/diagnostics13050903. PMID 36900047
- [Background] Moilanen M, Pirila E, Grenman R, Sorsa T, Salo T. Expression and regulation of collagenase-2 (MMP-8) in head and neck squamous cell carcinomas. J Pathol. 2002 May;197(1):72-81. doi: 10.1002/path.1078. PMID 12081207
- [Background] Guarnieri R, Zanza A, D'Angelo M, Di Nardo D, Del Giudice A, Mazzoni A, Reda R, Testarelli L. Correlation between Peri-Implant Marginal Bone Loss Progression and Peri-Implant Sulcular Fluid Levels of Metalloproteinase-8. J Pers Med. 2022 Jan 6;12(1):58. doi: 10.3390/jpm12010058. PMID 35055373
- [Background] Tchetverikov I, Ronday HK, Van El B, Kiers GH, Verzijl N, TeKoppele JM, Huizinga TW, DeGroot J, Hanemaaijer R. MMP profile in paired serum and synovial fluid samples of patients with rheumatoid arthritis. Ann Rheum Dis. 2004 Jul;63(7):881-3. doi: 10.1136/ard.2003.013243. PMID 15194590
- [Background] Weiss SJ. Tissue destruction by neutrophils. N Engl J Med. 1989 Feb 9;320(6):365-76. doi: 10.1056/NEJM198902093200606. No abstract available. PMID 2536474
- [Background] Feng Y, Li Q, Chen J, Yi P, Xu X, Fan Y, Cui B, Yu Y, Li X, Du Y, Chen Q, Zhang L, Jiang J, Zhou X, Zhang P. Salivary protease spectrum biomarkers of oral cancer. Int J Oral Sci. 2019 Jan 3;11(1):7. doi: 10.1038/s41368-018-0032-z. PMID 30602733
- [Background] Deng K, Pelekos G, Jin L, Tonetti MS. Diagnostic accuracy of a point-of-care aMMP-8 test in the discrimination of periodontal health and disease. J Clin Periodontol. 2021 Aug;48(8):1051-1065. doi: 10.1111/jcpe.13485. Epub 2021 Jun 10. PMID 33998040
- [Background] Bossuyt PM, Reitsma JB, Bruns DE, Gatsonis CA, Glasziou PP, Irwig L, Lijmer JG, Moher D, Rennie D, de Vet HC, Kressel HY, Rifai N, Golub RM, Altman DG, Hooft L, Korevaar DA, Cohen JF; STARD Group. STARD 2015: an updated list of essential items for reporting diagnostic accuracy studies. BMJ. 2015 Oct 28;351:h5527. doi: 10.1136/bmj.h5527. PMID 26511519
- [Background] Amin MB, Greene FL, Edge SB, Compton CC, Gershenwald JE, Brookland RK, Meyer L, Gress DM, Byrd DR, Winchester DP. The Eighth Edition AJCC Cancer Staging Manual: Continuing to build a bridge from a population-based to a more "personalized" approach to cancer staging. CA Cancer J Clin. 2017 Mar;67(2):93-99. doi: 10.3322/caac.21388. Epub 2017 Jan 17. PMID 28094848
- [Background] Preshaw PM, Hefti AF, Jepsen S, Etienne D, Walker C, Bradshaw MH. Subantimicrobial dose doxycycline as adjunctive treatment for periodontitis. A review. J Clin Periodontol. 2004 Sep;31(9):697-707. doi: 10.1111/j.1600-051X.2004.00558.x. PMID 15312090
- [Background] Maruyama Y, Nishimoto Y, Umezawa K, Kawamata R, Ichiba Y, Tsutsumi K, Kimura M, Murakami S, Kakizawa Y, Kumagai T, Yamada T, Fukuda S. Comparison of oral metabolome profiles of stimulated saliva, unstimulated saliva, and mouth-rinsed water. Sci Rep. 2022 Jan 13;12(1):689. doi: 10.1038/s41598-021-04612-x. PMID 35027617
- [Background] Drouin L, Overall CM, Sodek J. Identification of matrix metalloendoproteinase inhibitor (TIMP) in human parotid and submandibular saliva: partial purification and characterization. J Periodontal Res. 1988 Nov;23(6):370-7. doi: 10.1111/j.1600-0765.1988.tb01615.x. No abstract available. PMID 2851041
- [Background] Hsiao YC, Chi LM, Chien KY, Chiang WF, Chen SF, Chuang YN, Lin SY, Wu CC, Chang YT, Chu LJ, Chen YT, Chia SL, Chien CY, Chang KP, Chang YS, Yu JS. Development of a Multiplexed Assay for Oral Cancer Candidate Biomarkers Using Peptide Immunoaffinity Enrichment and Targeted Mass Spectrometry. Mol Cell Proteomics. 2017 Oct;16(10):1829-1849. doi: 10.1074/mcp.RA117.000147. Epub 2017 Aug 18. PMID 28821604
- [Background] Monea M, Pop AM. The Use of Salivary Levels of Matrix Metalloproteinases as an Adjuvant Method in the Early Diagnosis of Oral Squamous Cell Carcinoma: A Narrative Literature Review. Curr Issues Mol Biol. 2022 Dec 12;44(12):6306-6322. doi: 10.3390/cimb44120430. PMID 36547091
- [Background] Sorsa T, Nwhator SO, Sakellari D, Grigoriadis A, Umeizudike KA, Brandt E, Keskin M, Tervahartiala T, Parnanen P, Gupta S, Mohindra R, Bostanci N, Buduneli N, Raisanen IT. aMMP-8 Oral Fluid PoC Test in Relation to Oral and Systemic Diseases. Front Oral Health. 2022 Jun 10;3:897115. doi: 10.3389/froh.2022.897115. eCollection 2022. PMID 35757444
- [Background] Costa PP, Trevisan GL, Macedo GO, Palioto DB, Souza SL, Grisi MF, Novaes AB Jr, Taba M Jr. Salivary interleukin-6, matrix metalloproteinase-8, and osteoprotegerin in patients with periodontitis and diabetes. J Periodontol. 2010 Mar;81(3):384-91. doi: 10.1902/jop.2009.090510. PMID 20192865
- [Background] Johnson N, Ebersole JL, Kryscio RJ, Danaher RJ, Dawson D 3rd, Al-Sabbagh M, Miller CS. Rapid assessment of salivary MMP-8 and periodontal disease using lateral flow immunoassay. Oral Dis. 2016 Oct;22(7):681-7. doi: 10.1111/odi.12521. Epub 2016 Jul 14. PMID 27273425
- [Background] Sorsa T, Alassiri S, Grigoriadis A, Raisanen IT, Parnanen P, Nwhator SO, Gieselmann DR, Sakellari D. Active MMP-8 (aMMP-8) as a Grading and Staging Biomarker in the Periodontitis Classification. Diagnostics (Basel). 2020 Jan 22;10(2):61. doi: 10.3390/diagnostics10020061. PMID 31979091
- [Background] Lake BD. Histochemical detection of the enzyme deficiency in blood films in Wolman's disease. J Clin Pathol. 1971 Oct;24(7):617-20. doi: 10.1136/jcp.24.7.617. PMID 5118828
- [Background] Ala-aho R, Kahari VM. Collagenases in cancer. Biochimie. 2005 Mar-Apr;87(3-4):273-86. doi: 10.1016/j.biochi.2004.12.009. PMID 15781314
- [Background] Juurikka K, Butler GS, Salo T, Nyberg P, Astrom P. The Role of MMP8 in Cancer: A Systematic Review. Int J Mol Sci. 2019 Sep 11;20(18):4506. doi: 10.3390/ijms20184506. PMID 31514474
- [Background] Klein T, Bischoff R. Physiology and pathophysiology of matrix metalloproteases. Amino Acids. 2011 Jul;41(2):271-90. doi: 10.1007/s00726-010-0689-x. Epub 2010 Jul 18. PMID 20640864
- [Background] Dejonckheere E, Vandenbroucke RE, Libert C. Matrix metalloproteinase8 has a central role in inflammatory disorders and cancer progression. Cytokine Growth Factor Rev. 2011 Apr;22(2):73-81. doi: 10.1016/j.cytogfr.2011.02.002. Epub 2011 Mar 8. PMID 21388856
- [Background] Chung PC, Chan TC. Association between periodontitis and all-cause and cancer mortality: retrospective elderly community cohort study. BMC Oral Health. 2020 Jun 9;20(1):168. doi: 10.1186/s12903-020-01156-w. PMID 32517780
- [Background] Romandini M, Baima G, Antonoglou G, Bueno J, Figuero E, Sanz M. Periodontitis, Edentulism, and Risk of Mortality: A Systematic Review with Meta-analyses. J Dent Res. 2021 Jan;100(1):37-49. doi: 10.1177/0022034520952401. Epub 2020 Aug 31. PMID 32866427
- [Background] Gopinath D, Kunnath Menon R, K Veettil S, George Botelho M, Johnson NW. Periodontal Diseases as Putative Risk Factors for Head and Neck Cancer: Systematic Review and Meta-Analysis. Cancers (Basel). 2020 Jul 14;12(7):1893. doi: 10.3390/cancers12071893. PMID 32674369
- [Background] Komlos G, Csurgay K, Horvath F, Pelyhe L, Nemeth Z. Periodontitis as a risk for oral cancer: a case-control study. BMC Oral Health. 2021 Dec 15;21(1):640. doi: 10.1186/s12903-021-01998-y. PMID 34911520
- [Background] Bourgeois D, Inquimbert C, Ottolenghi L, Carrouel F. Periodontal Pathogens as Risk Factors of Cardiovascular Diseases, Diabetes, Rheumatoid Arthritis, Cancer, and Chronic Obstructive Pulmonary Disease-Is There Cause for Consideration? Microorganisms. 2019 Oct 9;7(10):424. doi: 10.3390/microorganisms7100424. PMID 31600905
- [Background] Rivera C. Essentials of oral cancer. Int J Clin Exp Pathol. 2015 Sep 1;8(9):11884-94. eCollection 2015. PMID 26617944
- [Background] Bosetti C, Carioli G, Santucci C, Bertuccio P, Gallus S, Garavello W, Negri E, La Vecchia C. Global trends in oral and pharyngeal cancer incidence and mortality. Int J Cancer. 2020 Aug 15;147(4):1040-1049. doi: 10.1002/ijc.32871. Epub 2020 Jan 30. PMID 31953840
- [Background] McIlwain WR, Sood AJ, Nguyen SA, Day TA. Initial symptoms in patients with HPV-positive and HPV-negative oropharyngeal cancer. JAMA Otolaryngol Head Neck Surg. 2014 May;140(5):441-7. doi: 10.1001/jamaoto.2014.141. PMID 24652023
- [Background] Guneri P, Epstein JB. Late stage diagnosis of oral cancer: components and possible solutions. Oral Oncol. 2014 Dec;50(12):1131-6. doi: 10.1016/j.oraloncology.2014.09.005. Epub 2014 Sep 23. PMID 25255960
- [Background] Cai M, Zheng Z, Bai Z, Ouyang K, Wu Q, Xu S, Huang L, Jiang Y, Wang L, Gao J, Pathak JL, Wu L. Overexpression of angiogenic factors and matrix metalloproteinases in the saliva of oral squamous cell carcinoma patients: potential non-invasive diagnostic and therapeutic biomarkers. BMC Cancer. 2022 May 11;22(1):530. doi: 10.1186/s12885-022-09630-0. PMID 35545767
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338